CLINICAL TRIAL: NCT06540378
Title: Stiripentol for the Treatment of Refractory Status Epilepticus
Status: Completed | Type: Observational
Sponsor: University Hospital Marburg (Other)
Responsible Party: Principal Investigator, Leona Möller, Leona Möller, MD; Principal Investigator, Consultant in Neurology, University Hospital Marburg
Other Study IDs: 24-61 RS
Record Dates: First submitted 2024-07-30; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Status Epilepticus
Keywords: Status epilepticus; Epilepsy; Stiripentol
MeSH Terms: conditions — Status Epilepticus; Epilepsy | interventions — stiripentol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- STP in RSE or SRSE: Patients received additional treatment of SE with STP
  Interventions: Drug: Stiripentol

INTERVENTIONS:
Drug: Stiripentol
  Other Names: Diacomit

SUMMARY:
The investigators retrospectively analyzed all patients who were admitted to the Department of Neurology at Marburg University Hospital between 2013 and 2023 with a diagnosis of (super)-refractory status epilepticus and who received additional treatment of SE with STP. All patients who received STP during the SE were included, regardless of previous medication.

DETAILED DESCRIPTION:
The investigators retrospectively analyzed all patients who were admitted to the Department of Neurology, University Hospital Marburg, Germany, between 2013 and 2023 with a diagnosis of status epilepticus, who received additional treatment of SE with STP. They were able to identify 25 patients who received STP as add on therapy. All these patients suffered from RSE or SRSE. Since there was no SOP or treatment algorithm available, they have listed the individual treatment regimens in Table 2. 5 of these patients were previously published in a case series (Strzelczyk et al. 2015).

Treatment success was defined as continuous interruption of the SE. Descriptive statistics are reported as absolute numbers and percentages, mean ± standard deviation (SD) or median ± median absolute deviation.

The study was approved by the local IRB.

ELIGIBILITY:
Inclusion Criteria:

* adult patients who suffered from RSE or SRSE and received STP as add on therapy.

Exclusion Criteria:

* children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators retrospectively analyzed all patients who were admitted to the Department of Neurology, University Hospital Marburg, Germany, between 2013 and 2023 with a diagnosis of status epilepticus, who received additional treatment of SE with STP. They were able to identify 25 patients who received STP as add on therapy. All these patients suffered from RSE or SRSE.
  Treatment success was defined as continuous interruption of the SE.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05 (Actual)

PRIMARY OUTCOMES:
Cessation of Status epilepticus | time to cessation of SE, normally during the first days of admission, up to one week
Number of participants with cessation of SE by STP | up to one week
Median dose of STP | From date of first admission until the date of first documented improvement of status epilepticus or severe sideeffects or termination due to lack of effect or date of death from any cause, whichever came first, assessed up to 12 months

SECONDARY OUTCOMES:
Treatment in combination with other anti-seizure medication | From date of first admission until the date of first documented improvement of status epilepticus or severe sideeffects or termination due to lack of effect or date of death from any cause, whichever came first, assessed up to 12 months
Individualised order of the anti-seizure medication administered | From date of first admission until the date of first documented improvement of status epilepticus or severe sideeffects or termination due to lack of effect or date of death from any cause, whichever came first, assessed up to 12 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moller L, Simon OJ, Junemann C, Austermann-Menche M, Bergmann MP, Habermehl L, Menzler K, Timmermann L, Strzelczyk A, Knake S. Stiripentol for the treatment of refractory status epilepticus. Neurol Res Pract. 2024 Oct 21;6(1):49. doi: 10.1186/s42466-024-00348-x. PMID 39428490